CLINICAL TRIAL: NCT00291330
Title: A Phase III, Randomised, Double Blind, Parallel-group Study of the Efficacy and Safety of Oral Dabigatran Etexilate 150 mg Twice Daily Compared to Warfarin (INR 2.0-3.0) for 6 Month Treatment of Acute Symptomatic Venous Thromboembolism (VTE), Following Initial Treatment (5-10 Days) With a Parenteral Anticoagulant Approved for This Indication.
Brief Title: Efficacy and Safety of Dabigatran Compared to Warfarin for 6 Month Treatment of Acute Symptomatic Venous Thromboembolism
Acronym: RE-COVER I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.53; 2005-001999-12 (EudraCT Number: EudraCT)
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-04

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Dabigatran; Warfarin

ARMS (2):
- dabigatran etexilate 150 mg (Experimental): twice daily
  Interventions: Drug: dabigatran etexilate 150 mg
- warfarin (INR 2-3) (Active Comparator): prn to maintain INR (2-3)
  Interventions: Drug: warfarin (INR 2-3)

INTERVENTIONS:
Drug: dabigatran etexilate 150 mg — twice daily
  Arms: dabigatran etexilate 150 mg
Drug: warfarin (INR 2-3) — prn to maintain INR (2-3)
  Arms: warfarin (INR 2-3)

SUMMARY:
The purpose of this trial is to determine the comparative safety and efficacy of dabigatran etexilate 150 mg bid administered orally and warfarin as needed (pro re nata - prn) to maintain an International Normalised Ratio (INR) of 2.0-3.0 for 6 month treatment of acute symptomatic venous thromboembolism (VTE), following initial treatment (5-10 days) with a parenteral anticoagulant approved for this indication. This trial aims to demonstrate non-inferiority of dabigatran compared with warfarin in patients with acute symptomatic VTE. After achieving non-inferiority, this trial also aims to establish superiority (by means of hierarchical tests) of dabigatran over warfarin.

ELIGIBILITY:
Inclusion criteria

1. Acute deep vein thrombosis (DVT) of the leg involving proximal veins, and/or pulmonary embolism (PE) iin patients for whom at least 6 months of anticoagulant therapy is considered appropriate
2. Male or female, being 18 years of age or older
3. Written informed consent for study participation

Exclusion criteria

1. Overt symptoms of VTE for longer than 2 weeks prior to enrolment
2. PE satisfying at least one of the following criteria: Haemodynamic instability, embolectomy is indicated or performed, thrombolytic therapy is indicated or performed, or suspected source of PE is other than the legs
3. Actual or anticipated use of vena cava filter
4. Contraindications to anticoagulant therapy
5. Patients who in the investigators opinion should not be treated with warfarin
6. Allergy to heparins or other alternate approved therapy used for initial treatment, warfarin or dabigatran, or to one of the excipients included in these medications
7. Patients who in the investigators judgement are perceived as having an excessive risk of bleeding
8. Known anaemia
9. Need of anticoagulant treatment for disorders other than VTE
10. Recent unstable cardiovascular disease
11. Elevated AST or ALT > 2x ULN
12. Liver disease expected to have any potential impact on survival
13. Patients who have developed transaminase elevations upon exposure to ximelagatran
14. Severe renal impairment
15. Women who are pregnant, nursing, or of childbearing potential who refuse to use a medically acceptable form of contraception
16. Participation in another clinical trial with an investigational drug during the last 30 days or previous participation in this study
17. Patients considered unsuitable for inclusion by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2564 (Actual)
Dates: Start 2006-02; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (250):
- United States (23):
  - 1160.53.01035 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1160.53.01056 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1160.53.01044 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.53.01033 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1160.53.01046 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1160.53.01019 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1160.53.01008 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1160.53.01010 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1160.53.01014 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.53.01023 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1160.53.01029 Boehringer Ingelheim Investigational Site, Pontiac, Michigan
  - 1160.53.01009 Boehringer Ingelheim Investigational Site, Saint Louis Park, Minnesota
  - 1160.53.01031 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 1160.53.01036 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1160.53.01025 Boehringer Ingelheim Investigational Site, Valhalla, New York
  - 1160.53.01027 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1160.53.01039 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1160.53.01030 Boehringer Ingelheim Investigational Site, Grand Forks, North Dakota
  - 1160.53.01013 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1160.53.01028 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1160.53.01052 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1160.53.01055 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
  - 1160.53.01017 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Argentina (6):
  - 1160.53.54017 Boehringer Ingelheim Investigational Site, Adrogué
  - 1160.53.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.53.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.53.54006 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.53.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1160.53.54010 Boehringer Ingelheim Investigational Site, Capital Federal
- Australia (6):
  - 1160.53.61002 Boehringer Ingelheim Investigational Site, Woolloongabba, Queensland
  - 1160.53.61004 Boehringer Ingelheim Investigational Site, Bedford Park, South Australia
  - 1160.53.61003 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.53.61001 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1160.53.61006 The Avenue Cardiovascular Centre, Windsor, Victoria
  - 1160.53.61005 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Austria (3):
  - 1160.53.43001 Boehringer Ingelheim Investigational Site, Graz
  - 1160.53.43003 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1160.53.43002 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (6):
  - 1160.53.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.53.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.53.32003 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.53.32007 Boehringer Ingelheim Investigational Site, Edegem
  - 1160.53.32005 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.53.32004 Boehringer Ingelheim Investigational Site, Liège
- Brazil (11):
  - 1160.53.55010 Boehringer Ingelheim Investigational Site, Brasília
  - 1160.53.55007 Boehringer Ingelheim Investigational Site, Campinas
  - 1160.53.55001 Boehringer Ingelheim Investigational Site, Cerqueira César - Sao Paulo
  - 1160.53.55002 Boehringer Ingelheim Investigational Site, Cerqueira César - São Paulo
  - 1160.53.55014 Boehringer Ingelheim Investigational Site, Cristo Rei - Curitiba
  - 1160.53.55011 Boehringer Ingelheim Investigational Site, Goiânia
  - 1160.53.55017 Boehringer Ingelheim Investigational Site, Paraná
  - 1160.53.55012 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1160.53.55016 Boehringer Ingelheim Investigational Site, Rio de Janeiro - RJ
  - 1160.53.55004 Boehringer Ingelheim Investigational Site, Santo André
  - 1160.53.55005 Boehringer Ingelheim Investigational Site, São José do Rio Preto
- Canada (18):
  - 1160.53.02006 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.53.02013 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.53.02021 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.53.02004 Boehringer Ingelheim Investigational Site, Saint Johns, New Brunswick
  - 1160.53.02001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.53.02002 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.53.02005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.53.02010 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.53.02022 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.53.02011 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1160.53.02015 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.53.02019 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.53.02008 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.53.02009 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.53.02014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.53.02017 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.53.02020 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1160.53.02003 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- Czechia (12):
  - 1160.53.42001 Boehringer Ingelheim Investigational Site, Brno
  - 1160.53.42002 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1160.53.42011 Boehringer Ingelheim Investigational Site, Hranice
  - 1160.53.42009 Boehringer Ingelheim Investigational Site, Jihlava
  - 1160.53.42012 Boehringer Ingelheim Investigational Site, Liberec
  - 1160.53.42015 Boehringer Ingelheim Investigational Site, Nový Jičín
  - 1160.53.42005 Boehringer Ingelheim Investigational Site, Ostrava-Vitkovice
  - 1160.53.42004 Boehringer Ingelheim Investigational Site, Prague
  - 1160.53.42014 Boehringer Ingelheim Investigational Site, Tábor
  - 1160.53.42016 Boehringer Ingelheim Investigational Site, Teplice
  - 1160.53.42010 Boehringer Ingelheim Investigational Site, Ústí nad Labem
  - 1160.53.42007 Boehringer Ingelheim Investigational Site, Zlín
- Denmark (6):
  - 1160.53.45008 Boehringer Ingelheim Investigational Site, Esbjerg
  - 1160.53.45009 Boehringer Ingelheim Investigational Site, Holbæk
  - 1160.53.45002 Boehringer Ingelheim Investigational Site, Kolding
  - 1160.53.45004 Boehringer Ingelheim Investigational Site, København NV
  - 1160.53.45007 Boehringer Ingelheim Investigational Site, København S
  - 1160.53.45006 Boehringer Ingelheim Investigational Site, Slagelse
- France (24):
  - 1160.53.3301A Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301B Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301C Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301D Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301E Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301F Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301H Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3301I Boehringer Ingelheim Investigational Site, Brest
  - 1160.53.3302A Boehringer Ingelheim Investigational Site, Lorient
  - 1160.53.3310A Boehringer Ingelheim Investigational Site, Montpellier
  - 1160.53.3310B Boehringer Ingelheim Investigational Site, Montpellier
  - 1160.53.3310C Boehringer Ingelheim Investigational Site, Montpellier
  - 1160.53.3308B Boehringer Ingelheim Investigational Site, Nancy
  - 1160.53.3303B Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.53.3303C Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.53.3303D Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.53.3303E Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.53.3303A Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
  - 1160.53.3311A Boehringer Ingelheim Investigational Site, Toulon Naval
  - 1160.53.3311B Boehringer Ingelheim Investigational Site, Toulon Naval
  - 1160.53.3311C Boehringer Ingelheim Investigational Site, Toulon Naval
  - 1160.53.3311D Boehringer Ingelheim Investigational Site, Toulon Naval
  - 1160.53.3311E Boehringer Ingelheim Investigational Site, Toulon Naval
  - 1160.53.3308A Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - 1160.53.49003 Boehringer Ingelheim Investigational Site, Cologne
  - 1160.53.49017 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.53.49018 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.53.49005 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.53.49007 Boehringer Ingelheim Investigational Site, München
  - 1160.53.49009 Boehringer Ingelheim Investigational Site, Püttlingen
- Greece (3):
  - 1160.53.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1160.53.30005 Boehringer Ingelheim Investigational Site, Athens
  - 1160.53.30006 Boehringer Ingelheim Investigational Site, Athens
- Hungary (9):
  - 1160.53.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.53.36006 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.53.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 1160.53.36013 Boehringer Ingelheim Investigational Site, Eger
  - 1160.53.36012 Boehringer Ingelheim Investigational Site, Gyula
  - 1160.53.36004 Boehringer Ingelheim Investigational Site, Miskolc
  - 1160.53.36003 Boehringer Ingelheim Investigational Site, Pécs
  - 1160.53.36010 Boehringer Ingelheim Investigational Site, Székesfehérvár
  - 1160.53.36011 Boehringer Ingelheim Investigational Site, Szombathely
- India (13):
  - 1160.53.91011 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.53.91012 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.53.91019 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.53.91013 Boehringer Ingelheim Investigational Site, Indore
  - 1160.53.91021 Boehringer Ingelheim Investigational Site, Karna
  - 1160.53.91022 Boehringer Ingelheim Investigational Site, Kerala
  - 1160.53.91020 Boehringer Ingelheim Investigational Site, Ludhiana
  - 1160.53.91007 Boehringer Ingelheim Investigational Site, Mysore
  - 1160.53.91015 Boehringer Ingelheim Investigational Site, Nagpur
  - 1160.53.91010 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.53.91005 Boehringer Ingelheim Investigational Site, Pune
  - 1160.53.91008 Boehringer Ingelheim Investigational Site, Pune
  - 1160.53.91004 Boehringer Ingelheim Investigational Site, Vadodara
- Israel (9):
  - 1160.53.97202 Boehringer Ingelheim Investigational Site, Afula
  - 1160.53.97207 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1160.53.97211 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.53.97203 Boehringer Ingelheim Investigational Site, Holon
  - 1160.53.97205 Boehringer Ingelheim Investigational Site, KfarSaba
  - 1160.53.97206 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1160.53.97210 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.53.97204 Boehringer Ingelheim Investigational Site, Tel Litwinsky
  - 1160.53.97201 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (6):
  - 1160.53.39003 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.53.39002 Boehringer Ingelheim Investigational Site, Padua
  - 1160.53.39001 Boehringer Ingelheim Investigational Site, Perugia
  - 1160.53.39004 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1160.53.39007 Boehringer Ingelheim Investigational Site, Vimercate
  - 1160.53.39005 Boehringer Ingelheim Investigational Site, Vittorio Veneto (tv)
- Mexico (3):
  - 1160.53.5264 Boehringer Ingelheim Investigational Site, Chihuahua City
  - 1160.53.5270 Boehringer Ingelheim Investigational Site, Culiacán
  - 1160.53.5262 Boehringer Ingelheim Investigational Site, San Luis Potosí City
- Netherlands (8):
  - 1160.53.31010 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.53.31001 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1160.53.31006 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.53.31013 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1160.53.31005 Boehringer Ingelheim Investigational Site, Maastricht
  - 1160.53.31002 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 1160.53.31004 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.53.31009 Boehringer Ingelheim Investigational Site, Rotterdam
- New Zealand (4):
  - 1160.53.64003 Boehringer Ingelheim Investigational Site, Auckland
  - 1160.53.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1160.53.64002 Boehringer Ingelheim Investigational Site, Otahuhu Auckland
  - 1160.53.64001 Boehringer Ingelheim Investigational Site, Takapuna Auckland
- Norway (4):
  - 1160.53.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.53.47004 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.53.47003 Boehringer Ingelheim Investigational Site, Rud
  - 1160.53.47005 Boehringer Ingelheim Investigational Site, Trondheim
- Portugal (5):
  - 1160.53.35104 Boehringer Ingelheim Investigational Site, Almada
  - 1160.53.35109 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.53.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.53.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 1160.53.35105 Boehringer Ingelheim Investigational Site, Lisbon
- Russia (17):
  - 1160.53.07011 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1160.53.07021 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1160.53.07016 Boehringer Ingelheim Investigational Site, Krasnodar
  - 1160.53.07004 Boehringer Ingelheim Investigational Site, Kursk
  - 1160.53.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.53.07010 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1160.53.07020 Boehringer Ingelheim Investigational Site, Omsk
  - 1160.53.07018 Boehringer Ingelheim Investigational Site, Pskov
  - 1160.53.07009 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.53.07023 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.53.07024 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.53.07025 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.53.07001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.53.07014 Boehringer Ingelheim Investigational Site, Ufa
  - 1160.53.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.53.07006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.53.07007 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (5):
  - 1160.53.42107 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1160.53.42106 Boehringer Ingelheim Investigational Site, Lučenec
  - 1160.53.42102 Boehringer Ingelheim Investigational Site, Nitra
  - 1160.53.42103 Boehringer Ingelheim Investigational Site, Nové Zámky
  - 1160.53.42104 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (9):
  - 1160.53.27007 Boehringer Ingelheim Investigational Site, Centurion
  - 1160.53.27001 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.53.27002 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.53.27004 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.53.27006 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.53.27009 Suite 404, Medical Centre, Pretoria
  - 1160.53.27003 Boehringer Ingelheim Investigational Site, Randburg
  - 1160.53.27008 Suite M5, Second Floor, Richards Bay
  - 1160.53.27005 Boehringer Ingelheim Investigational Site, Roodepoort
- Spain (10):
  - 1160.53.34012 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1160.53.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.53.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.53.34007 Boehringer Ingelheim Investigational Site, Cartagena. Murcia
  - 1160.53.34003 Boehringer Ingelheim Investigational Site, Cuenca
  - 1160.53.34009 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.53.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.53.34004 Boehringer Ingelheim Investigational Site, Santander
  - 1160.53.34005 Boehringer Ingelheim Investigational Site, Torrelavega.Santander
  - 1160.53.34011 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (7):
  - 1160.53.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.53.46006 Boehringer Ingelheim Investigational Site, Jönköping
  - 1160.53.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.53.46007 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.53.46008 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.53.46005 Boehringer Ingelheim Investigational Site, Sundsvall
  - 1160.53.46003 Boehringer Ingelheim Investigational Site, Uppsala
- Turkey (Türkiye) (7):
  - 1160.53.90003 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.53.90004 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.53.90005 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.53.90001 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.53.90002 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.53.90007 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.53.90006 Boehringer Ingelheim Investigational Site, Izmir
- Ukraine (3):
  - 1160.53.38006 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.53.38005 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1160.53.38003 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (7):
  - 1160.53.44008 Boehringer Ingelheim Investigational Site, Aberdeen
  - 1160.53.44005 Boehringer Ingelheim Investigational Site, Headington, Oxford
  - 1160.53.44004 Boehringer Ingelheim Investigational Site, London
  - 1160.53.44009 Boehringer Ingelheim Investigational Site, London
  - 1160.53.44011 Boehringer Ingelheim Investigational Site, London
  - 1160.53.44006 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1160.53.44012 Boehringer Ingelheim Investigational Site, Sheffield

REFERENCES:
- [Derived] Goldhaber SZ, Eriksson H, Kakkar A, Schellong S, Feuring M, Fraessdorf M, Kreuzer J, Schueler E, Schulman S. Efficacy of dabigatran versus warfarin in patients with acute venous thromboembolism in the presence of thrombophilia: Findings from RE-COVER(R), RE-COVER II, and RE-MEDY. Vasc Med. 2016 Dec;21(6):506-514. doi: 10.1177/1358863X16668588. Epub 2016 Nov 1. PMID 27807306
- [Derived] Schulman S, Kakkar AK, Goldhaber SZ, Schellong S, Eriksson H, Mismetti P, Christiansen AV, Friedman J, Le Maulf F, Peter N, Kearon C; RE-COVER II Trial Investigators. Treatment of acute venous thromboembolism with dabigatran or warfarin and pooled analysis. Circulation. 2014 Feb 18;129(7):764-72. doi: 10.1161/CIRCULATIONAHA.113.004450. Epub 2013 Dec 16. PMID 24344086
- [Derived] Majeed A, Hwang HG, Connolly SJ, Eikelboom JW, Ezekowitz MD, Wallentin L, Brueckmann M, Fraessdorf M, Yusuf S, Schulman S. Management and outcomes of major bleeding during treatment with dabigatran or warfarin. Circulation. 2013 Nov 19;128(21):2325-32. doi: 10.1161/CIRCULATIONAHA.113.002332. Epub 2013 Sep 30. PMID 24081972
- [Derived] Schulman S, Kearon C, Kakkar AK, Mismetti P, Schellong S, Eriksson H, Baanstra D, Schnee J, Goldhaber SZ; RE-COVER Study Group. Dabigatran versus warfarin in the treatment of acute venous thromboembolism. N Engl J Med. 2009 Dec 10;361(24):2342-52. doi: 10.1056/NEJMoa0906598. PMID 19966341
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1160/1160.53_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2564 patients enrolled/randomised in this trial but only 2539 started treatment
Groups:
- Dabigatran 150 mg: bid (twice daily) oral
- Warfarin: PRN to maintain an INR of 2.0-3.0
Period: Overall Study
Arm/Group | Dabigatran 150 mg | Warfarin
Started | 1273 (Started Treatment) | 1266 (Started Treatment)
Completed | 1172 (Completed planned observation time) | 1169 (Completed planned observation time)
Not Completed | 101 | 97
Not completed — Adverse Event | 47 | 40
Not completed — Protocol Violation | 13 | 20
Not completed — Lost to Follow-up | 16 | 11
Not completed — Withdrawal by Subject | 22 | 25
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 150 mg | Warfarin | Total
Number analyzed (Participants) | 1273 | 1266 | 2539
Age, Continuous [Mean (Standard Deviation); unit: Year] | 55.0 (15.8) | 54.4 (16.2) | 54.7 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 535 | 520 | 1055
  Male | 738 | 746 | 1484
Acute symptomatic DVT of the leg and/or PE as assessed by investigator [Number; unit: participants] — Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE)
  participants
    Symptomatic PE and symptomatic DVT | 121 | 124 | 245
    Symptomatic PE | 270 | 271 | 541
    Symptomatic DVT | 880 | 869 | 1749
    No PE and no DVT | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Symptomatic Venous Thromboembolism (VTE) and Deaths Related to VTE
Description: All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: For statistical analysis 1: from randomisation to end of post treatment period (ptp), planned to be up to day 224. For statistical analysis 2: from randomisation to 6 months (up to day 180)
Population: Full analysis set (FAS): consisted of all randomised patients who were documented to have taken at least one dose of study drug. Patients were assigned to the treatment groups as randomised, i.e. regardless of the actual medication taken.
Measure: Number; unit: Participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
Participants
  Participants with event (up to day 180) | 30 | 27
  Participants with event (up to end of ptp) | 34 | 32
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio vs. Warfarin (events occurring between randomisation and end of post treatment period). The time to first occurrence of the primary endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Non-Inferiority or Equivalence — Non inferiority margin was set up to 2.75 for the HR analysis; p < 0.0001, Regression, Cox — Non-inferiority P-Value. Two Statistical analyses performed on primary endpoint. Both non inferiority for the risk difference and for the hazard ratio analyses to be reached in order to conclude positively on the primary endpoint; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 1.05, 95% CI [0.65 to 1.70]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference vs. Warfarin for Proportion of patients with VTE or death related to VTE at 6 months. Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Non-Inferiority or Equivalence — Non inferiority margin was set up to 3.6% for the risk difference based on KM estimates; p < 0.0001, Kaplan Meier weighted estimates — [p-value comment as in outcome 1, analysis 1]; Risk Difference (Percentage) = 0.40, 95% CI [-0.80 to 1.50]
Statistical Analysis 3: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio vs. Warfarin (events occurring between randomisation and the day 180). The time to first occurrence of the primary endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; Regression, Cox; Patients without events are censored at day 180; Hazard Ratio (HR) = 1.10, 95% CI [0.65 to 1.84]

2. Secondary Outcome: Number of Participants With Recurrent Symptomatic VTE and All Deaths
Description: VTE or any death which occured from randomisation to end of post treatment period.
  All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: For statistical analysis 1: from randomisation to 6 months (up to day 180) For statistical analysis 2: from randomisation to end of ptp, planned to be up to day 224.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
Participants
  Participants with event (up to day 180) | 48 | 44
  Participants with event (up to end of ptp) | 55 | 53
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference vs. Warfarin for Proportion of patients with VTE or death at 6 months. Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.6220, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.30, 95% CI [-1.00 to 1.70]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio vs. Warfarin (events occurring between randomisation and end of post treatment period). The time to first occurrence of the endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; p = 0.9844, Regression, Cox; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 1.00, 95% CI [0.69 to 1.46]

3. Secondary Outcome: Number of Participants With Recurrent Symptomatic DVT
Description: Symptomatic DVT which occured from randomisation to end of post treatment period.
  All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
participants
  Participants with event (up to day 180) | 16 | 18
  Participants with event (up to end of ptp) | 17 | 22
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference vs. Warfarin for Proportion of patients with symptomatic DVT at 6 months. Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.6466, Kaplan Meier weighted estimates; Risk Difference (Percentage) = -0.20, 95% CI [-1.10 to 0.70]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3850, Regression, Cox; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 0.76, 95% CI [0.40 to 1.42]

4. Secondary Outcome: Number of Participants With Recurrent Symptomatic Non-fatal PE
Description: Symptomatic non-fatal PE which occured from randomisation to end of post treatment period.
  All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
participants
  Participants with event (up to day 180) | 13 | 7
  Participants with event (up to end of ptp) | 16 | 8
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference vs. Warfarin for Proportion of patients with symptomatic non-fatal PE at 6 months. Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.2981, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.30, 95% CI [-0.30 to 1.00]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1092, Regression, Cox; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 2.00, 95% CI [0.86 to 4.68]

5. Secondary Outcome: Number of Participants Who Died Due to VTE
Description: VTE - related deaths which occured from randomisation to end of post treatment period.
  All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
participants
  Participants with event (up to day 180) | 1 | 3
  Participants with event (up to end of ptp) | 1 | 3
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference at 6 months vs. Warfarin for Proportion of patients who died due to VTE . Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.5327, Kaplan Meier weighted estimates; Risk Difference (Percentage) = -0.30, 95% CI [-1.20 to 0.60]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3332, Regression, Cox; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 0.33, 95% CI [0.03 to 3.15]

6. Secondary Outcome: Number of Participants Who Died (Any Cause)
Description: Any deaths which occured from randomisation to end of post treatment period. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1274 | 1265
participants
  Participants with event (up to day 180) | 21 | 21
  Participants with event (up to end of ptp) | 25 | 25
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Risk difference at 6 months vs. Warfarin for Proportion of patients who died from any cause. Point estimate and 95% CI for the overall risk difference obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.8018, Kaplan Meier weighted estimates; Risk Difference (Percentage) = -0.10, 95% CI [-1.00 to 0.80]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.8203, Regression, Cox; Patients without events are censored at the end of post treatment period (day 224); Hazard Ratio (HR) = 0.94, 95% CI [0.54 to 1.63]

7. Secondary Outcome: Number of Participants With Bleeding Events
Description: Major bleeding events (MBE) were defined as
  * Fatal bleeding
  * Symptomatic bleeding in a critical area or organ
  * Bleeding causing a fall in haemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of 2 or more units of whole blood or red cells
  Clinically-relevant bleeding events (CRBE) was defined as
  * spontaneous skin hematoma >=25 cm²
  * spontaneous nose bleed >5 min
  * macroscopic hematuria spontaneous or >24 hours if associated with an intervention
  * spontaneous rectal bleeding (more than spotting on toilet paper)
  * gingival bleeding >5 min
  * leading to hospitalisation and / or requiring surgical treatment
  * leading to a transfusion of <2 units of whole blood or red cells
  * any other bleeding event considered clinically relevant by the investigator
  Any bleeding events were defined as major, clinically-relevant and nuisance bleeding events. Nuisance bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: From first intake of study drug to last intake of study drug + 6 days washout (washout time can be reduced until 0 day if the patient takes an other anti-coagulant therapy on and after last intake of active study drug)
Population: Treated set (TS): consisted of all randomised patients who were documented to have taken at least one dose of study drug. Patients were assigned to the treatment groups as treated.
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1273 | 1266
participants
  Major bleeding events | 20 | 24
  MBE and/or CRBE | 71 | 111
  Any bleeding events | 207 | 280
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio vs. Warfarin for the category major bleeding events (events occurring between 1st intake of study drug and last intake of study drug + 6 days). The time to first occurrence of the endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; p = 0.5063, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI [0.45 to 1.48]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio vs. Warfarin for the category of any bleeding events (events occurring between 1st intake of study drug and last intake of study drug + 6 days). The time to first occurrence of the endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.59 to 0.85]

8. Secondary Outcome: Number of Participants With Acute Coronary Syndrome (ACS)
Description: Any ACS occurring during the conduct of the study (centrally adjudicated as definite).
  Counts of patients having a centrally adjudicated definite ACS during intake of active study drug, after stopping active study drug and before or without intake of active study drug, according to treatment group.
  All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: From first intake of study drug to end of study conduct
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1273 | 1266
participants
  During intake of active study drug | 5 | 3
  After stopping active study drug | 4 | 2
  Before/without intake of active study drug | 2 | 0

9. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1204 | 1198
participants
  AST increase | 21 | 22
  AST decrease | 0 | 0
  ALT increase | 26 | 38
  ALT decrease | 0 | 0
  Bilirubin increase | 7 | 13
  Bilirubin decrease | 0 | 0

ADVERSE EVENTS:
Time Frame: From first intake of study drug to last intake of study drug + 6 days washout (washout time can be reduced until 0 day if the patient takes an other anti-coagulant therapy on and after last intake of active study drug)
Arm/Group | Dabigatran 150 mg | Warfarin
Serious Adverse Events (participants affected / at risk) | 165/1273 | 150/1266
Other Adverse Events (participants affected / at risk) | 163/1273 | 209/1266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 150 mg (N=1273) | Warfarin (N=1266)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal symptom (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 6 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 4 | 6
Death (General disorders) | 1 | 1
Drug ineffective (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Haemorrhagic cyst (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 4
Polyp (General disorders) | 1 | 0
Pseudocyst (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 3
Empyema (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 5 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 8
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Biopsy bladder (Investigations) | 0 | 1
Cardiac imaging procedure abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Investigation (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1
Troponin I increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute polyneuropathy (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 9
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Bartholinitis (Reproductive system and breast disorders) | 1 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 10 | 9
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Iliac artery thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 150 mg (N=1273) | Warfarin (N=1266)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 63 | 69
Headache (Nervous system disorders) | 78 | 87
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.